CLINICAL TRIAL: NCT02251340
Title: Randomized Controlled Trial of an Eczema Care Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Corinna Rea, Staff Physician, Instructor in Medicine, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChildrensH
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Eczema
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Families in the intervention group will receive an Eczema Care Plan
  Interventions: Behavioral: Eczema Care Plan
- Control (No Intervention): Families in the control group will not receive an Eczema Care Plan

INTERVENTIONS:
Behavioral: Eczema Care Plan
  Arms: Intervention

SUMMARY:
The objectives of this project are to increase families' understanding of eczema and improve eczema management in the primary care setting. We have created an "Eczema Care Plan" similar to those used in the management of asthma. It gives specific instructions about medications, bathing and moisturizing, as well as when to seek further treatment. We will conduct a randomized controlled trial of the plan in Primary Care at Longwood for a 10 month period. Specifically, we aim to (1) decrease eczema severity (2) improve patient quality of life and (3) increase parental knowledge and confidence about eczema management. We also plan to track provider uptake and documentation of the plan and elicit feedback from parents and providers on the utility and feasibility of the plan.

ELIGIBILITY:
Inclusion Criteria:a) accompanying adult speaks English b) patient has a history of eczema c) patient is between the ages of 1 month and 16 years d) family is coming for an eczema visit or plans to discuss eczema e) accompanying adult is a primary caregiver f) child is not in foster care g) caregiver has not received an eczema care plan previously. -

Exclusion Criteria: a) accompanying adult does not speak English b) patient does not have a history of eczema c) patient is younger than 1 month or older than 16 years of age d) eczema will not be discussed at the visit e) accompanying adult is not the primary caregiver f) child is in foster care g) caregiver has received an eczema care plan previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
proportion of patients with moderate/severe/very severe eczema | 1 month for each patient
quality of life measured via validated survey | 1 month for each patient
parental knowledge measured via survey | 1 month for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States